CLINICAL TRIAL: NCT04375267
Title: Phase I Trial With 177Lu-DOTA-TATE and Olaparib in Somatostatin Receptor Positive Tumours
Brief Title: 177Lu-DOTA-TATE and Olaparib in Somatostatin Receptor Positive Tumours
Acronym: LuPARP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001700-37
Record Dates: First submitted 2020-04-27; First posted 2020-05-05 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Clinical Trial, Phase I; Neuroendocrine Tumors; Thymoma; Mesothelioma
MeSH Terms: conditions — Neuroendocrine Tumors; Thymoma; Mesothelioma | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-DOTA-TATE and olaparib (Experimental)
  Interventions: Drug: 177Lu-DOTA-TATE + olaparib

INTERVENTIONS:
Drug: 177Lu-DOTA-TATE + olaparib — 177Lu-DOTA-TATE in four cycles in combination with escalated doses of olaparib

SUMMARY:
This is a phase I study of 177Lu-DOTA-TATE in combination with the PARP-inhibitor olaparib for treatment of patients with somatostatin receptor positive tumours detected by 68Ga-DOTA-TATE/TOC PET. The combination of a PARP inhibitor that will specifically target the repair mechanism, with ionising radiation causing SSB's might overcome the repair dependent survival of the tumour cells, making them more sensitive to β-emission and increase the probability of tumour cell death.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of neoplasia (not mandatory for meningioma)
* GEPNETs grade 3 or aggressive grade 2 tumours with a poor prognosis and a Ki67 > 15% OR neuroendocrine tumours NOS after standard therapy OR thymomas/tumours of other origin after standard therapy OR meningiomas after standard therapy not suitable for surgery or radiotherapy
* Evidence of regional or distant metastases or localised disease not accessible for complete resection
* Measurable disease according to RECIST 1.1
* Evidence of somatostatin receptor positive disease detected by 68Ga-DOTA-TATE/TOC PET
* Progressive disease during the last 14 months based on CT or new lesions detected by 68Ga-DOTA-TATE PET.
* Performance status ECOG 0 - 1
* Life expectancy > 6 months
* Age >18 years, no upper age limit.
* Neutrophil count >1,5 x 109/L
* Platelet count >100 x 109/L
* Normal liver function regarding transaminases, PK and albumin. A raised bilirubin which can be considered an isolated effect of liver metastases is not a contraindication as long as the levels remain <1.5 x ULN.
* GFR > 50 ml/min
* Written informed consent from patients
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Exclusion Criteria:

* Performance Status ECOG > 1
* Well differentiated GEPNETs grad 1 and 2 (except aggressive grade 2 tumours with a poor prognosis and a Ki67 > 15%)
* Loco-regional treatment during the last 3 months involving all of the measurable lesions
* Chemotherapy during the last 8 weeks or longer until no persisting toxicity exists. Earlier treatment with mTORi or TKI the last 4 weeks or until no persisting toxicity exists
* Previous treatment with 177Lu-DOTA-TATE or cis-/carboplatin
* Other concomitant nephrotoxic treatment
* Serious heart disease (NYHA III-IV)
* Previous radiotherapy including >25% of active bone marrow volume
* Pregnancy and lactation
* Extensive liver metastases combined with impaired liver function (i.e. abnormal laboratory parameters (> grad 1 CTCAE) or ascites)
* Symptomatic CNS metastases (e.g. requiring corticosteroid treatment) Symptomatic treatment for meningiomas or corticosteroids due to treatment related swelling is however allowed
* Ongoing treatment with interferon. This treatment should be suspended a minimum of 4 wees before treatment with 177Lu-DOTA-TATE, or longer if there is persisting signs of toxicity
* Patients who have a another metastatic tumor diagnosis
* Known or expected hypersensitivity to 177Lu-DOTA-TATE, 68Ga- DOTA-TATE/TOC or any of their excipients
* History of psychiatric disease/condition that may interfere with the objectives and assessments of the study
* Female subjects who are pregnant or breastfeeding or subjects of reproductive potential who are not willing to employ effective birth control methods (Pearl index <1) from screening to 6 months after the last dose of olaparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 6 months after last treatment cycle
  To assess the number of participants with toxicity of 177Lu-DOTA-TATE in combination with olaparib measured by NCI Common Toxicity Criteria v 5.0

SECONDARY OUTCOMES:
TTP | 3 years
  Time to progression
Response rate | 12 months after last treatment cycle
  Response rate (RECIST) at 3 and 12 months
OS | 3 years
  Overall survival
DOR | 3 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Oncology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hallqvist A, Svensson J, Hagmarker L, Marin I, Ryden T, Beauregard JM, Bernhardt P. Optimizing the Schedule of PARP Inhibitors in Combination with 177Lu-DOTATATE: A Dosimetry Rationale. Biomedicines. 2021 Oct 29;9(11):1570. doi: 10.3390/biomedicines9111570. PMID 34829796